CLINICAL TRIAL: NCT04758247
Title: Evaluation of the TheraNova Neuromodulation System for the Treatment of Overactive Bladder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD-10-1330
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: TheraNova Neuromodulation System
- Sham (Sham Comparator)
  Interventions: Device: TheraNova Neuromodulation System

INTERVENTIONS:
Device: TheraNova Neuromodulation System — The investigational device is a transcutaneous electrical nerve stimulation (TENS) device that is designed to provide stimulation to the nerves at the site of application via surface electrodes temporarily adhered to the skin.

SUMMARY:
To evaluate the safety and effectiveness of the TheraNova Neuromodulation System in overactive bladder (OAB) patients. The primary safety endpoint will be device-related adverse events. The primary effectiveness endpoint will be urinary urge incontinence (UUI) responder rate at 12 weeks (a responder is defined as a subject who experiences at least a 50% reduction in the mean frequency of UUI events per day from baseline to 12 weeks as measured in the 3-day voiding diaries). Responder rate will be compared between subjects randomized to the active treatment vs. the sham treatment.

ELIGIBILITY:
Inclusion Criteria:

Women and men ≥18 years of age

* Individual has a diagnosis of OAB with urge urinary incontinence or mixed incontinence (urge and stress) with urge urinary incontinence being the most bothersome type of urinary incontinence for at least 6 months (self-reported)
* Individual has ≥4 incontinence events with associated moderate or severe urgency (UUI events), with at least one UUI event per day, as recorded in the baseline 3-day voiding diary
* Individual has a mean frequency of urinary voiding events per day ≥10 times in one 24-hour day as recorded in the baseline 3-day voiding diary
* Individual is ambulatory and able to use the toilet independently
* Individual has not taken antimuscarinics, anticholinergics or beta-3 agonists for at least 2 weeks prior to enrollment
* Individual is able to provide informed consent
* Individual is capable and willing to follow all study-related procedures

Exclusion Criteria:

* • Individual has stress urinary incontinence as the most bothersome type of urinary incontinence (self-report)

  * Individual has an abnormal post-void residual urine volume (>150 cc at baseline)
  * Male who has a clinically significant bladder outlet obstruction (assessed by uroflow, maximum flow rate <15 mL/s for a voided volume of at least 150 cc)
  * Male who has been previously diagnosed with Benign Prostate Hyperplasia
  * Male who has abnormal serum PSA (>2.5 ng/mL)
  * Individual has abnormal serum creatinine levels (>1.2 mg/dL for women and >1.4 mg/dL for men)
  * Individual has history of chronic kidney disease
  * Female of childbearing age (≤50 years old) who is pregnant as confirmed by urine pregnancy test, or who plans to become pregnant during the study period
  * Female who is less than one-year post-partum and/or is breast-feeding
  * Female with a clinically significant pelvic organ prolapse (≥ stage III on POP-Q evaluation)
  * Individual has diabetes with peripheral nerve compromise or severe uncontrolled diabetes (HbA1C ≥ 8.5)
  * Individual has known polyuria
  * Individual has an active urinary tract infection (UTI) at the time of enrollment
  * Individual has recurrent UTI defined as ≥4 UTIs in the past 12 months
  * Individual has peripheral arterial disease
  * Individual has the presence of a urinary fistula, bladder stone, or interstitial cystitis
  * Individual has a diagnosis of prostate, urethral, or bladder cancer
  * Individual has morbid obesity (BMI ≥ 40)
  * Individual has clinically significant urethral stricture disease or bladder neck contracture
  * Individual has a metallic implant that is exposed above the bone surface (e.g. a bone fracture fixation plate, but not an embedded bone screw) and is located under the skin on the bottom of the foot for either or under the skin on the anterior aspect of the mid-thigh for either leg.
  * Individual has an implanted electrical and/or neurostimulator device (e.g. pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
  * Individual has had previous treatment with sacral neuromodulation
  * Individual has been treated with percutaneous tibial nerve stimulation or pelvic floor muscle stimulation
  * Individual is currently using, or has used in the past 3 months, transcutaneous electrical nerve stimulation (TENS) in the pelvic region, back, legs, or feet
  * Individual has been treated with onabotulinumtoxinA in the past 9 months
  * Individual has a clinically significant peripheral neuropathy
  * Individual has a history of pelvic pain as primary diagnosis in the past 12 months (VAS score of >4 (scale of 0 to 10))
  * Individual has neurogenic bladder (i.e. Multiple Sclerosis, Parkinson's, Spinal Cord Injury)
  * Individual has used an investigational drug, biologic, or medical device in the past 4 weeks
  * Individual is deemed unsuitable for enrollment in the study by the investigator based on the subject's history or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness endpoint is the percentage of subjects with at least a 50% reduction in frequency of UUI events from baseline to 12 weeks as measured in 3-day voiding diaries. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC Davis Health, Sacramento, California
  - Stanford Medicine, Stanford, California